CLINICAL TRIAL: NCT05886621
Title: Pilot RCT to Test the Integrated mHealth App Intervention (SiS-H) for Smoking Cessation for People With HIV
Brief Title: Testing the Integrated mHealth App Intervention "SiS-H"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Bettina B. Hoeppner, Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023P001360; R21CA261458 (NIH)
Record Dates: First submitted 2023-05-23; First posted 2023-06-02 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2024-09

CONDITIONS: Smoking Cessation
Keywords: smoking; smartphone app; smoking cessation; QuitGuide; Smiling instead of Smoking; SiS-H; positive psychology; mHealth; QUIT; Life Steps
MeSH Terms: conditions — Smoking Cessation; Smoking

STUDY DESIGN:
Intervention Model Description: 2-group pilot randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smiling instead of Smoking - HIV (Experimental): Participants will be onboarded to the smartphone app "Smiling instead of Smoking - HIV" (SiS-H), and will be asked to use it for 8 weeks while they quit smoking.
  Interventions: Behavioral: Smiling instead of Smoking - HIV
- QuitGuide (Active Comparator): Participants will be onboarded to the smartphone app "QuitGuide" (QG), and will be asked to use it for 8 weeks while they quit smoking.
  Interventions: Behavioral: QuitGuide

INTERVENTIONS:
Behavioral: Smiling instead of Smoking - HIV — Participants will be onboarded to the smartphone app "Smiling instead of Smoking - HIV" (SiS-H) and will be asked to complete the integrated SiS-H program while they quit smoking. The integrated SiS-H treatment consists of: (1) face-to-face onboarding to the SiS-H app, (2) one face-to-face session discussing app usage and antiretroviral therapy (ART) adherence (Life Steps), with direct linkage to tools in the app supporting ART adherence, and (3) an 8-week course of the SiS-H app. The SiS-H app is a smoking cessation app that uses a positive psychology framework in conjunction with with the US Clinical Practice Guidelines for smoking cessation to guide participants through the process of quitting smoking.
  Other Names: SiS-H
  Arms: Smiling instead of Smoking - HIV
Behavioral: QuitGuide — Participants will be onboarded to the NCI smartphone app QuitGuide(QG) and will be asked to use it for 8 weeks to support them in quitting smoking. The QuitGuide app follows the US Clinical Practice Guidelines. The app is freely available on NCI's Smokefree.gov website, which is a recommended resource for treating smokers in the healthcare setting. The QuitGuide app is frequently used as a comparison app in smartphone app smoking cessation studies. It asks participants to set a quit day, track their mood and cravings, and log their cigarettes. It provides app users with guidance on quitting (i.e., "Learn to Quit" information), offers strategies to counter smoking triggers, and allows users to set reminders to stay smoke free (time and location based).
  Other Names: QG
  Arms: QuitGuide

SUMMARY:
The present study is a pilot randomized controlled trial (RCT) that seeks to test the feasibility, acceptability, process outcomes, and exploratory outcomes of a newly integrated, app-based smoking cessation treatment (SiS-H, which stands for "Smiling instead of Smoking for people with HIV") for people with HIV who smoke. This treatment will be compared to onboarding to the National Cancer Institute's smartphone app "QuitGuide" (QG). Persons with HIV who smoke and are engaged in HIV clinical care (n=64) will be randomized (1:1) to smoking cessation support via SiS-H vs. "QuitGuide".

DETAILED DESCRIPTION:
The team recently developed an mHealth intervention that integrates (1) the "Smiling instead of Smoking" (SiS) app, a conceptually-grounded, iteratively developed smoking cessation smartphone app, (2) a successful face-to-face smoking cessation treatment for smokers with HIV, called QUIT, and (3) Life Steps, an efficacious brief intervention to promote adaptive engagement in HIV care. The new integrated treatment emphasizes protecting the experience of positive emotions among smokers with HIV as they navigate the process of quitting smoking and supports smoking self-efficacy by engaging participants in app-based activities. Guidance and support for engaging with the app are provided through two face-to-face sessions.

The present study is a pilot randomized controlled trial (RCT) that seeks to test the feasibility, acceptability, process outcomes and exploratory outcomes of this new treatment, called SiS-H, compared to onboarding to the National Cancer Institute's smartphone app "QuitGuide" (QG). Smokers with HIV engaged in HIV clinical care (n=64) will be randomized (1:1) to smoking cessation support via SiS-H vs. the National Cancer Institute's smartphone app "QuitGuide" (QG).

Smoking cessation support will last 8 weeks and will consist of face-to-face interactions with study staff about navigating their assigned smoking cessation app and brief smoking cessation information. Participants will be offered nicotine replacement patches but will not be required to use them.

Study assessments will consist of online surveys (baseline, 2, 6, and 12 weeks post-quit), and biochemical tests of smoking status (baseline, 12 weeks post-quit). Data will be extracted from the medical record, with participants' permission.

The aims of the study are:

1. To test the feasibility and acceptability of the SiS-H integrated treatment to support people with HIV in quitting smoking.
2. To test the efficacy of the integrated SiS-H treatment to have a positive impact on variables relevant to the process of quitting smoking.
3. (EXPLORATORY) To examine differences in 30-day point prevalence smoking abstinence (biologically verified), other smoking outcomes, and HIV medication adherence between both app groups.

Below are specifics on the Specific Aims of this study, and the investigators' hypotheses:

Specific Aim 1: In this pilot randomized-controlled trial, the investigators will test the feasibility and acceptability of the SiS-H integrated treatment to support people with HIV in quitting smoking.

1. Feasibility (primary outcome): App use of the assigned app, as measured by the number of days participants used the app during the treatment period (8 weeks) will be significantly higher in SiS-H compared to QG. App use will be calculated based on passively collected app usage data.
2. Feasibility (secondary outcomes): The investigators hypothesize that SiS-H treatment will be feasible, as measured in the following ways:

   1. Self-reported time spent applying content; the investigators' hypothesis is that "time spent" (i.e., as measured by this self-report item: "During the past week, how much time did participants spend applying or contemplating the content of the [Smiling Instead of Smoking app / QuitGuide app (logic-branched by treatment group)]? ______________ (in minutes, total for the week)") will be equal or higher in SiS-H than QG
   2. Achieving expected app use (i.e., 75% of participants using the app at least once 6 out of 8 weeks of the prescribed treatment week)
   3. Use of smoking cessation strategies (see attached instrument); the investigators' hypothesis is that "use of strategies" will be equal or higher in SiS-H than QG
3. Acceptability (secondary outcomes): The investigators hypothesize that SiS-H treatment will be acceptable (i.e., equal or higher scores compared to the control group), as measured at treatment end in the following ways:

   1. Satisfaction with smoking cessation support (Client Satisfaction Questionnaire (CSQ-8))
   2. App system usability (System Usability Scale (SUS))
   3. User app rating (User Mobile Application Rating Scale (uMARS))

Specific Aim 2: In this pilot RCT, the investigators will test the efficacy of the integrated SiS-H treatment to have a positive impact on variables relevant to the process of quitting smoking. Specifically, the investigators hypothesize outcomes will be better for the SiS-H group compared to the QG group at the end of treatment on the following measures:

1. Smoking cessation self-efficacy as measured by the Smoking Self-Efficacy Questionnaire (SEQ-12); higher self-efficacy is considered 'better'
2. Craving, as measured by the Brief Questionnaire of Smoking Urges (QSU-Brief); lower craving is considered 'better'
3. Positive affect, as measured by the positive affect subscale of the PANAS Positive and Negative Affect Schedule (PANAS); higher positive affect is considered 'better'

Exploratory Aim 3: Although not statistically powered, the investigators will examine differences in 30-day point prevalence abstinence (biologically verified), other smoking outcomes, and 30-day self-reported ART adherence, as measured by the Medication Adherence scale, between both app groups.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years of age
* current smoker, who has smoked at least 100 cigarettes lifetime, and smokes at least weekly
* HIV positive, by self-report
* currently engaged in HIV clinical care (i.e., saw an HIV care provider within the last year)
* willing to let study staff look at medical record to extract HIV-relevant information (e.g., CD4 T cell count)
* willing to make a quit attempt as part of this study
* willing to give permission to study staff to look at app usage for the assigned smoking cessation app
* willing and able to comply with study procedures

Exclusion Criteria:

* does not own a smartphone
* does not have daily access to the owned smartphone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2023-11-07 (Actual); Primary Completion 2025-05-05 (Actual); Study Completion 2025-07-07 (Actual)

PRIMARY OUTCOMES:
App usage | Continuously logged in the app from baseline (2 weeks pre-quit) to end of treatment (6 weeks post-quit).
  Number of days participants used the assigned app during the prescribed period of app use (i.e., 8 weeks for both apps). App usage is passively recorded by the app, which time-stamps every interaction with the app.

SECONDARY OUTCOMES:
Time spent applying content | Measured at week 4 (2 weeks post-quit) and week 8 (6-weeks post-quit)
  Time spent applying content will be measured with the self-report item: "During the past week, how much time did you spend applying or contemplating the content of the [Smiling Instead of Smoking app / QuitGuide app (logic-branched by treatment group)]? ______________ (in minutes, total for the week)").
Expected app usage | Assessed at end of treatment (6 weeks post-quit)
  A percentage based on the categorical re-coding of the actual app usage, measured in days, where YES indicates that participants used the app at least once during 6 out of the 8 weeks of the prescribed treatment weeks, and NO indicates that participants used the app less often.
Use of smoking cessation strategies | Assessed at end of treatment (6 weeks post-quit)
  Assessed using an 8-item measure in which participants rate the extent to which they agree or disagree with statements about the smoking cessation support they received and the things they did while quitting (5-point Likert scale, 1=strongly disagree, 5=strongly agree, e.g., "I used techniques to help me relax"). Higher scores indicate greater use of smoking cessation strategies.
Satisfaction with smoking cessation support | Assessed at end of treatment (6 weeks post-quit)
  As measured using the Client Satisfaction Scale (CSQ-8), an 8 item multiple choice measure that will be used to assess participants' satisfaction with the smoking cessation support they receive (e.g., "How satisfied are you with the amount of help you received?"). Scores are summed across items and range from 8 to 32, with higher scores indicating greater satisfaction.
App usability rating, System Usability Scale (SUS) | Assessed at end of treatment (6 weeks post-quit)
  As assessed via the System Usability Scale (SUS), a ten-item attitude scale giving a global view of subjective assessments of usability, adapted to include language specific to the smoking app (e.g., "I found the smoking app unnecessarily complex" 5-point Likert: 1 = strongly disagree, 5 = strongly agree). Scale scores range from 0 to 100 with greater scores indicating a more favorable perception of usability of the app.
User mobile application rating (uMARS) | Assessed at end of treatment (6 weeks post-quit)
  User app ratings will be assessed using the Mobile Application Rating Scale user version (uMARS). The uMARS is a self-report form with 26 items that assess participant's evaluations of various app features. Dimensions of this measure include engagement (5 items), functionality (4 items), aesthetics (3 items), information quality (4 items), app subjectivity quality (4 items), and perceived impact (6 items). Items are rated on differently worded 5-point Likert scales ranging from 1 (Inadequate) to 5 (Excellent). An overall app rating score can be calculated as the mean score of the first 16 questions (range of 1-5), with higher scores meaning higher overall perceived app quality.
Smoking Self-Efficacy Questionnaire (SEQ-12) | Measured at baseline, week 4 (2 weeks post-quit), week 8 (6-weeks post-quit)
  The Smoking Self-Efficacy Questionnaire (SEQ-12) is a two-dimensional 12-item self-report scale measuring a person's confidence in his or her ability to abstain from smoking when facing internal stimuli (e.g. feeling depressed) and external stimuli (e.g. being with smokers) on a 0-100 slider scale (i.e., 0=not at all confident that I can refrain; 100=extremely confident that I can refrain). Scale scores are created by mean scoring across items and range from 0 to 100. Higher scores indicate greater self-efficacy to abstain from smoking.
Positive affect - Positive and Negative Affect Schedule (PANAS) | Measured at baseline, week 4 (2 weeks post-quit), week 8 (6-weeks post-quit)
  Positive affect will be measured using the Positive and Negative Affect Schedule (PANAS). This 20-item scale asks participants to indicate how they felt in the past week, using a 5-point Likert scale ranging from 1="very slightly or not at all" to 5="extremely." Scores for 10 positive words and 10 negative words will be summed separately and will be reported as mean scores (not scale totals) ranging from 1-5, with lower scores indicating low (positive or negative) affect and higher scores indicating high (positive or negative) affect. The 10 items for POSITIVE (PA) affect are attentive, interested, alert, excited, enthusiastic, inspired, proud, determined, strong, and active.
Negative affect - Positive and Negative Affect Schedule (PANAS) | Measured at baseline, week 4 (2 weeks post-quit), week 8 (6-weeks post-quit)
  Negative affect will be measured using the Positive and Negative Affect Schedule (PANAS). This 20-item scale asks participants to indicate how they felt in the past week, using a 5-point Likert scale ranging from 1="very slightly or not at all" to 5="extremely." Scores for 10 positive words and 10 negative words will be summed separately and will be reported as mean scores (not scale totals) ranging from 1-5, with lower scores indicating low (positive or negative) affect and higher scores indicating high (positive or negative) affect. The 10 items for NEGATIVE (NA) affect are distressed, upset, hostile, irritable, scared, afraid, ashamed, guilty, nervous, and jittery.
Brief Questionnaire of Smoking Urges (QSU) | Measured at baseline, week 4 (2 weeks post-quit), week 8 (6-weeks post-quit)
  Smoking urges will be assessed using the Questionnaire of Smoking Urges. This 10-item scale assesses overall nicotine dependence, craving, and smoking withdrawal symptoms. Items will be rated on a 7-point Likert-scale ranging from 1=Strongly disagree to 7=Strongly agree. We will present the mean instead of total scores for ease in interpretation, so that scale scores can range from 1.0 to 7.0, with higher scores indicating greater smoking urges.
Attitudes Towards Smoking Scale (ATS) - adverse effects of smoking sub-scale | Measured at baseline, week 4 (2 weeks post-quit), week 8 (6-weeks post-quit)
  Smoking attitudes will be assessed using the Attitudes Towards Smoking Scale (ATS-18). The 18-item self-report ATS-18 measures attitudes towards smoking in current and former cigarette smokers. It is rated on a 5-point Likert scale, from 1="strongly disagree" to 5="strongly agree.". The ATS-18 has 3 sub-scales: Adverse effects of smoking (items 1-10), psychoactive benefits of smoking (items 11-14), and pleasure of smoking (items 15-18). To score, all items per sub-scale will be averaged to obtain a mean score within each sub-scale. For each sub-scale, higher scores indicate greater agreement with the specific attitude towards smoking.
Attitudes Towards Smoking Scale (ATS) - psychoactive benefits of smoking sub-scale | Measured at baseline, week 4 (2 weeks post-quit), week 8 (6-weeks post-quit)
  Smoking attitudes will be assessed using the Attitudes Towards Smoking Scale (ATS-18). The 18-item self-report ATS-18 measures attitudes towards smoking in current and former cigarette smokers. It is rated on a 5-point Likert scale, from 1="strongly disagree" to 5="strongly agree.". The ATS-18 has 3 sub-scales: Adverse effects of smoking (items 1-10), psychoactive benefits of smoking (items 11-14), and pleasure of smoking (items 15-18). To score, all items per sub-scale will be averaged to obtain a mean score within each sub-scale. For each sub-scale, higher scores indicate greater agreement with the specific attitude towards smoking.
Attitudes Towards Smoking Scale (ATS) - pleasure of smoking sub-scale | Measured at baseline, week 4 (2 weeks post-quit), week 8 (6-weeks post-quit)
  Smoking attitudes will be assessed using the Attitudes Towards Smoking Scale (ATS-18). The 18-item self-report ATS-18 measures attitudes towards smoking in current and former cigarette smokers. It is rated on a 5-point Likert scale, from 1="strongly disagree" to 5="strongly agree.". The ATS-18 has 3 sub-scales: Adverse effects of smoking (items 1-10), psychoactive benefits of smoking (items 11-14), and pleasure of smoking (items 15-18). To score, all items per sub-scale will be averaged to obtain a mean score within each sub-scale. For each sub-scale, higher scores indicate greater agreement with the specific attitude towards smoking.
Decisional Balance Inventory (DBI) for Smoking - negative expectancies sub-scale | Measured at baseline, week 4 (2 weeks post-quit), week 8 (6-weeks post-quit)
  Negative smoking expectancies will be assessed using the Decisional Balance Inventory (DBI) for Smoking Short Form. This 6-item form assesses the personal importance people place on positive and negative smoking expectancies. Items are rated on slider scales ranging from 0="not at all important" to 100="extremely important." Two sub-scale mean scores will be calculated: positive expectancies (3 items), and negative smoking expectancies (3 items). On both scales, higher scores indicate a greater importance of the smoking expectancies (positive or negative).
Decisional Balance Inventory (DBI) for Smoking - positive expectancies subscale | Measured at baseline, week 4 (2 weeks post-quit), week 8 (6-weeks post-quit)
  Positive smoking expectancies will be assessed using the Decisional Balance Inventory (DBI) for Smoking Short Form. This 6-item form assesses the personal importance people place on positive and negative smoking expectancies. Items are rated on slider scales ranging from 0="not at all important" to 100="extremely important." Two sub-scale mean scores will be calculated: positive expectancies (3 items), and negative smoking expectancies (3 items). On both scales, higher scores indicate a greater importance of the smoking expectancies (positive or negative).
Modified version of the Twenty Statements Test | Measured at baseline, week 4 (2 weeks post-quit), week 8 (6-weeks post-quit)
  The depth of the thought-action repertoire will be assessed using a modified version of the Open-Ended Twenty Statements Test (MOETST). The original MOETST usually starts by evoking an emotion, asks participants to name the emotion they experienced and keep it in mind, and then list all the things they would like to do 'right now'. Instead of using emotion inductions, we will ask participants to think of their upcoming quit date (at baseline) or when last using their assigned app treatment, and then fill out as many action statements as they can think of (limited to a maximum of 20) with the prompt "Instead of smoking at that moment, I could have ....". The number of actions will be summed to produce a though-action repertoire score with a range of 0-20, with higher scores indicating a richer thought-action repertoire.

OTHER OUTCOMES:
30-day point prevalence abstinence (PPA) - self-reported | Measured at baseline, week 4 (2 weeks post-quit), week 8 (6-weeks post-quit)
  Participants will be asked to report whether they were abstinent some cigarette smoking during the last 30 days (yes vs. no). Missing data will be interpreted as smoking.
30-day point prevalence abstinence (PPA) - biochemically verified | Measured at baseline and week 20 (3 months after end of treatment)
  Participants will provide breath samples for expired carbon monoxide (CO; cutoff value of < 5 ppm). For CO-confirmed stated abstinence of 7 days or longer, abstinence will be verified by saliva cotinine using the NicAlert or similar test strip (based on availability; we will use test strips detecting 30ng of cotinine, where the test strip will indicate 'smoking' if the saliva content exceeds 30ng). This information will be combined with the self-reported abstinence data; reports of smoking abstinence that conflict with biochemical verification will be overridden with smoking status YES.
HIV Medication Adherence | Measured at baseline, week 4 (2 weeks post-quit), week 8 (6-weeks post-quit)
  HIV medication will be assessed with a 3-item medication adherence questionnaire. The three items ask about the number of days on which participants missed doses, the number of days when participants did not take medication as directed, and how well they followed directions. The answer options will be linearly transformed to 0-100 scales, averaged, and will generate a score between 0 and 100, with 0 being the lowest adherence and 100 being the highest adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Hoeppner, PhD, MS, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Behavioral Medicine Program (BMED), Boston, Massachusetts, United States

REFERENCES:
- [Background] Brooke, J. (1996). SUS: A 'quick and dirty' usability scale. In P. W. Jordan, B. Thomas, I. L. McClelland, & B. Weerdmeester (Eds.), Usability evaluation in industry (1st ed., Vol. 189, pp. 4-7). CRC Press.
- [Background] Cox LS, Tiffany ST, Christen AG. Evaluation of the brief questionnaire of smoking urges (QSU-brief) in laboratory and clinical settings. Nicotine Tob Res. 2001 Feb;3(1):7-16. doi: 10.1080/14622200020032051. PMID 11260806
- [Background] Etter JF, Bergman MM, Humair JP, Perneger TV. Development and validation of a scale measuring self-efficacy of current and former smokers. Addiction. 2000 Jun;95(6):901-13. doi: 10.1046/j.1360-0443.2000.9569017.x. PMID 10946439
- [Background] Etter JF, Humair JP, Bergman MM, Perneger TV. Development and validation of the Attitudes Towards Smoking Scale (ATS-18). Addiction. 2000 Apr;95(4):613-25. doi: 10.1046/j.1360-0443.2000.95461312.x. PMID 10829336
- [Background] Fredrickson BL, Branigan C. Positive emotions broaden the scope of attention and thought-action repertoires. Cogn Emot. 2005 May 1;19(3):313-332. doi: 10.1080/02699930441000238. PMID 21852891
- [Background] Larsen DL, Attkisson CC, Hargreaves WA, Nguyen TD. Assessment of client/patient satisfaction: development of a general scale. Eval Program Plann. 1979;2(3):197-207. doi: 10.1016/0149-7189(79)90094-6. No abstract available. PMID 10245370
- [Background] Stoyanov SR, Hides L, Kavanagh DJ, Wilson H. Development and Validation of the User Version of the Mobile Application Rating Scale (uMARS). JMIR Mhealth Uhealth. 2016 Jun 10;4(2):e72. doi: 10.2196/mhealth.5849. PMID 27287964
- [Background] Ward RM, Velicer WF, Rossi JS, Fava JL, Prochaska JO. Factorial invariance and internal consistency for the decisional balance inventory--short form. Addict Behav. 2004 Jul;29(5):953-8. doi: 10.1016/j.addbeh.2004.02.042. PMID 15219341
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Wilson IB, Lee Y, Michaud J, Fowler FJ Jr, Rogers WH. Validation of a New Three-Item Self-Report Measure for Medication Adherence. AIDS Behav. 2016 Nov;20(11):2700-2708. doi: 10.1007/s10461-016-1406-x. PMID 27098408

DOCUMENTS (1):
  • Informed Consent Form (2024-11-08): https://cdn.clinicaltrials.gov/large-docs/21/NCT05886621/ICF_000.pdf